CLINICAL TRIAL: NCT02624973
Title: PErsonalized TREatment of High-risk MAmmary Cancer - the PETREMAC Trial
Acronym: PETREMAC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Vest (Other); Pfizer (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015/8463
Record Dates: First submitted 2015-11-30; First posted 2015-12-09 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: neoadjuvant treatment; personalized medicine
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin; palbociclib; Cyclophosphamide; Trastuzumab; pertuzumab; olaparib; Mastectomy, Segmental; Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- A (Experimental): ER/PGR>50% TP53 wt
  Interventions: Drug: Neoadjuvant tamoxifen + goserelin (premenopausal women); Drug: Neoadjuvant letrozole (postmenopausal women); Drug: Neoadjuvant endocrine therapy + palbociclib (if lack of response to endocrine therapy alone); Procedure: Breast conserving surgery or mastectomy + SNB/axillary dissection; Radiation: Postoperative radiotherapy breast/chest wall + regional lymph nodes; Drug: Adjuvant letrozole (postmenopausal women); Drug: Adjuvant tamoxifen + goserelin (premenopausal women); Drug: Adjuvant palbociclib (if palbociclib given neoadjuvant); Drug: Adjuvant Epirubicin+ Cyclophosphamide
- B (Experimental): ER/PGR>50% TP53 mutated
  Interventions: Drug: Neoadjuvant docetaxel + cyclophosphamide; Procedure: Breast conserving surgery or mastectomy + SNB/axillary dissection; Radiation: Postoperative radiotherapy breast/chest wall + regional lymph nodes; Drug: Adjuvant letrozole (postmenopausal women); Drug: Adjuvant tamoxifen + goserelin (premenopausal women)
- C (Experimental): ER/PGR<50% TP53 wt
  Interventions: Drug: Neoadjuvant docetaxel; Procedure: Breast conserving surgery or mastectomy + SNB/axillary dissection; Radiation: Postoperative radiotherapy breast/chest wall + regional lymph nodes; Drug: Adjuvant letrozole (postmenopausal women); Drug: Adjuvant tamoxifen + goserelin (premenopausal women)
- D (Experimental): ER/PGR<50% TP53 mutated
  Interventions: Drug: Neoadjuvant docetaxel + cyclophosphamide; Procedure: Breast conserving surgery or mastectomy + SNB/axillary dissection; Radiation: Postoperative radiotherapy breast/chest wall + regional lymph nodes; Drug: Adjuvant letrozole (postmenopausal women); Drug: Adjuvant tamoxifen + goserelin (premenopausal women)
- E (Experimental): HER2+ TP53 wt
  Interventions: Drug: Neoadjuvant docetaxel + trastuzumab + pertuzumab; Procedure: Breast conserving surgery or mastectomy + SNB/axillary dissection; Radiation: Postoperative radiotherapy breast/chest wall + regional lymph nodes; Drug: Adjuvant trastuzumab; Drug: Adjuvant letrozole (postmenopausal women); Drug: Adjuvant tamoxifen + goserelin (premenopausal women)
- F (Experimental): HER2+ TP53 mutated
  Interventions: Drug: Neoadjuvant docetaxel + cyclophosphamide + trastuzumab + pertuzumab; Procedure: Breast conserving surgery or mastectomy + SNB/axillary dissection; Radiation: Postoperative radiotherapy breast/chest wall + regional lymph nodes; Drug: Adjuvant trastuzumab; Drug: Adjuvant letrozole (postmenopausal women); Drug: Adjuvant tamoxifen + goserelin (premenopausal women)
- G (Experimental): Triple negative breast cancer TP53 wt
  Interventions: Drug: Neoadjuvant olaparib; Drug: Neoadjuvant cyclophosphamide (after 10 weeks of olaparib alone); Procedure: Breast conserving surgery or mastectomy + SNB/axillary dissection; Radiation: Postoperative radiotherapy breast/chest wall + regional lymph nodes
- H (Experimental): Triple negative breast cancer TP53 mutated
  Interventions: Drug: Neoadjuvant olaparib; Drug: Neoadjuvant cyclophosphamide (after 10 weeks of olaparib alone); Procedure: Breast conserving surgery or mastectomy + SNB/axillary dissection; Radiation: Postoperative radiotherapy breast/chest wall + regional lymph nodes

INTERVENTIONS:
Drug: Neoadjuvant tamoxifen + goserelin (premenopausal women)
  Arms: A
Drug: Neoadjuvant letrozole (postmenopausal women)
  Arms: A
Drug: Neoadjuvant endocrine therapy + palbociclib (if lack of response to endocrine therapy alone)
  Arms: A
Drug: Neoadjuvant docetaxel + cyclophosphamide
  Arms: B; D
Drug: Neoadjuvant docetaxel
  Arms: C
Drug: Neoadjuvant docetaxel + trastuzumab + pertuzumab
  Arms: E
Drug: Neoadjuvant docetaxel + cyclophosphamide + trastuzumab + pertuzumab
  Arms: F
Drug: Neoadjuvant olaparib
  Arms: G; H
Drug: Neoadjuvant cyclophosphamide (after 10 weeks of olaparib alone)
  Arms: G; H
Procedure: Breast conserving surgery or mastectomy + SNB/axillary dissection — After response to neoadjuvant treatment
Radiation: Postoperative radiotherapy breast/chest wall + regional lymph nodes
Drug: Adjuvant trastuzumab
  Arms: E; F
Drug: Adjuvant letrozole (postmenopausal women)
  Arms: A; B; C; D; E; F
Drug: Adjuvant tamoxifen + goserelin (premenopausal women)
  Arms: A; B; C; D; E; F
Drug: Adjuvant palbociclib (if palbociclib given neoadjuvant)
  Arms: A
Drug: Adjuvant Epirubicin+ Cyclophosphamide
  Arms: A

SUMMARY:
Breast cancer is an optimal "model disease" for studying personalized medicine. Breast cancer was the first malignancy for which a predictive factor forecasting response to therapy was identified nearly 50 years ago; the expression of the estrogen receptor (ER). Furthermore, breast cancer is by far the malignancy in which prognostic and predictive factors have been most extensively studied. Primary medical treatment (pre-surgical medical therapy) offers a unique setting to explore predictive factors due to the fact that primary breast cancers are easily accessible to repeated tissue sampling and evaluation of therapy response both clinically and radiologically. For many years, the investigators have studied predictive factors in primary medical treatment of breast cancer. In the present project, the investigators will implement a new trial concept where the current knowledge from previous trials with respect to predictive markers (hormone receptors, HER2; TP53, CHEK2 and RB1), will be combined with massive parallel sequencing (MPS). Thereby, the investigators aim to design the "next-generation" primary medical treatment where 1) therapy regimens are individualized based on a limited number of known predictive factors and, 2) MPS is used to explore additional predictive factors and their co-regulators in order to fully identify the mechanisms of drug sensitivity / resistance across individual tumours and pave the way for further personalized breast cancer therapy in the future. As for the new era of "genomic medicine", the current trial concept will allow individual tumours to be characterized by their unique gene mutation / epigenetic modification profile upfront, to allocate patients to their optimal personalized medicine as compared to "classical" drug testing through phase II/III trials.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histologically confirmed non-inflammatory breast cancer, >4 cm in diameter and /or metastatic ipsilateral axillary deposits for which the smallest diameter of the largest node >2 cm by CT or ultrasound scan.
* WHO performance status 0-1
* Known tumor ER, PGR, HER2 and TP53 status.
* Known tumor Ki67 percentage (if ER/PGR>50% and TP53 wt status).
* Distant metastasis not suspected. Patients will undergo radiology exams during screening phase, after signing the informed consent.
* Age >18 years
* Patients must have clinically and/or radiographically documented measurable breast cancer according to RECIST.
* Radiology studies (CT thorax/abdomen and bone scintigraphy/bone scan) must be performed within 28 days prior to registration.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration/randomization, written informed consent must be given according to national and local regulations.
* For arms B-H:

  * Neutrophils > 1.5 x 109/L
  * Platelets > 100 x 109/L
  * Bilirubin < 2 x upper limit normal (ULN). For patients with Gilbert´s syndrome bilirubin >2 x ULN is accepted if there is no evidence of biliary obstruction.
  * Serum creatinine < 1.5 x ULN
  * ALT and Alk Phos (ALP) <2.5 x ULN
  * INR < 1.5

Exclusion Criteria:

* Unstable angina pectoris or heart failure
* Other co-morbidity that, based on the assessment of the treating physician, may preclude the use of chemotherapy at actual doses.
* Pregnant or lactating patients can not be included.
* Clinical evidence of serious coagulopathy. Prior arterial/venous thrombosis or embolism does not exclude patients from inclusion, unless patient is considered unfit by study oncologist.
* Patient not able to give an informed consent or comply with study regulations as deemed by study investigator.
* Active cystitis (to be treated upfront)
* Active bacterial infections
* Urinary obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Predictive and prognostic value of mutations in 300 cancer-related genes assessed in breast cancer tissue by next generation sequencing before starting neoadjuvant therapy. | Ten years
  Primary endpoint

SECONDARY OUTCOMES:
To assess genetic/epigenetic changes within the tumor tissue during therapy | Before vs. 16-24 wks after treatment start. Four years: summary of all patients treated.
  Secondary endpoint
The objective response rate (ORR) of personalized medicine, compared to ORR for best standard-of-care using historical data for comparison | Four years
  Secondary endpoint
Tumor Ki67 reduction after 2 and 5 weeks of treatment in Arm A | Assessment for each patient after 2 and 5 weeks of treatment. Four years - summary of all patients in arm A.
  Secondary endpoint
To estimate recurrence-free and overall survival when patients are treated with the optimal personalized treatment available as of 2015, using historical data for comparison | Ten years
  Secondary endpoint
To evaluate the percentage of patients completing neoadjuvant treatment and completing surgery | Four years
  Secondary endpoint
Breast conserving surgery rate (potential to avoid mastectomy) | Four years
  Secondary endpoint
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Ten years
  Secondary endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Hans Petter Eikesdal, MD PhD, Principal Investigator — Consultant oncologist
Locations (7):
- Norway (7):
  - Akershus University Hospital, Lørenskog, Akershus
  - Haukeland University Hospital, Bergen, Hordaland
  - Helse Fonna, Haugesund, Rogaland
  - Helse Stavanger, Stavanger, Rogaland
  - Helse Førde, Førde, Sogn Og Fjordande
  - St. Olavs Hospital, Trondheim, Sør Trøndelag
  - Helse Nord/UNN, Tromsø, Troms

IPD SHARING:
Plan to Share IPD: Yes
Tumor genomic data will be made available after publication.

REFERENCES:
- [Result] Eikesdal HP, Yndestad S, Elzawahry A, Llop-Guevara A, Gilje B, Blix ES, Espelid H, Lundgren S, Geisler J, Vagstad G, Venizelos A, Minsaas L, Leirvaag B, Gudlaugsson EG, Vintermyr OK, Aase HS, Aas T, Balmana J, Serra V, Janssen EAM, Knappskog S, Lonning PE. Olaparib monotherapy as primary treatment in unselected triple negative breast cancer. Ann Oncol. 2021 Feb;32(2):240-249. doi: 10.1016/j.annonc.2020.11.009. Epub 2020 Nov 24. PMID 33242536
- [Derived] Yndestad S, Engebrethsen C, Herencia-Ropero A, Nikolaienko O, Vintermyr OK, Lillestol RK, Minsaas L, Leirvaag B, Iversen GT, Gilje B, Blix ES, Espelid H, Lundgren S, Geisler J, Aase HS, Aas T, Gudlaugsson EG, Llop-Guevara A, Serra V, Janssen EAM, Lonning PE, Knappskog S, Eikesdal HP. Homologous Recombination Deficiency Across Subtypes of Primary Breast Cancer. JCO Precis Oncol. 2023 Sep;7:e2300338. doi: 10.1200/PO.23.00338. PMID 38039432
- [Derived] Wang L, Wang D, Sonzogni O, Ke S, Wang Q, Thavamani A, Batalini F, Stopka SA, Regan MS, Vandal S, Tian S, Pinto J, Cyr AM, Bret-Mounet VC, Baquer G, Eikesdal HP, Yuan M, Asara JM, Heng YJ, Bai P, Agar NYR, Wulf GM. PARP-inhibition reprograms macrophages toward an anti-tumor phenotype. Cell Rep. 2022 Oct 11;41(2):111462. doi: 10.1016/j.celrep.2022.111462. PMID 36223740
- [Derived] Batalini F, Gulhan DC, Mao V, Tran A, Polak M, Xiong N, Tayob N, Tung NM, Winer EP, Mayer EL, Knappskog S, Lonning PE, Matulonis UA, Konstantinopoulos PA, Solit DB, Won H, Eikesdal HP, Park PJ, Wulf GM. Mutational Signature 3 Detected from Clinical Panel Sequencing is Associated with Responses to Olaparib in Breast and Ovarian Cancers. Clin Cancer Res. 2022 Nov 1;28(21):4714-4723. doi: 10.1158/1078-0432.CCR-22-0749. PMID 36048535